CLINICAL TRIAL: NCT06172192
Title: EFFECTS OF CORE STRENGTHENING WITH RESISTIVE VERSUS NON-RESISTIVE DIAPHRAGMATIC TRAINING ON CORE ENDURANCE IN LOWER CROSS SYNDROME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/23
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Lower Cross Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A will perform Core Strengthening exercises. In addition to core strengthening protocol, non-resistive Diaphragmatic training group will perform self-diaphragm breathing exercises
  Core strengthening protocol will comprise of following three phases:
  1. Warm up phase:
  2. Core strengthening phase:
  3. Cool down phase:
  After performance of Core Strengthening protocol, Group A will perform Self-Diaphragmatic breathing exercises.
  Interventions: Procedure: Core Strengthening; Procedure: Self-Diaphragm breathing exercises
- Group B (Experimental): Group B will perform Core Strengthening exercises. In addition to core strengthening protocol, resistive Diaphragmatic training group will perform resisted-diaphragm breathing exercises.
  Core strengthening protocol will comprise of following three phases:
  1. Warm up phase
  2. Core strengthening phase
  3. Cool down phase
  After performance of Core Strengthening protocol, group B will perform Resistive Diaphragmatic Exercises.
  Interventions: Procedure: Core Strengthening; Procedure: Resistive-Diaphragm breathing exercises

INTERVENTIONS:
Procedure: Core Strengthening — 1. Warm up phase Following exercise would be performed in warm up. Jump rope, Cross jacks, Standing side crunch, Mountain climbers, Scissor skier, Criss cross crunches, Reverse lunge high kick, Inchworm, Hip circles, Bent over.
  2. Core Strengthening:
     Abdominal bracing, Bracing with heel slides, Bracing with leg lifts, Bracing with bridging, Bracing in standing, Bracing with standing row exercise, Quadruped arm lifts with bracing, Quadruped leg lifts with bracing, Quadruped alternate arm and leg lifts with bracing , Oblique abdominals
  3. Cool down phase: Following exercise would be performed for cood down: child pose, Ab stretch, cat cow stretch, hip stretch, oblique stretch, standing forward bend.
  After performance of core strengthening protocol, group A will perform self-diaphragmatic breathing exercises while group B will perform resistive diaphragmatic breathing exercise.
Procedure: Self-Diaphragm breathing exercises — Participants will place one hand on the chest and other on the abdomen, feeling the swelling of the stomach and the movement of the chest. It will be performed in supine position.
  Supervised breathing exercises in two sets for 15 minutes with 5 minutes break between sets and 10 minutes rest after it will be performed
  Arms: Group A
Procedure: Resistive-Diaphragm breathing exercises — Participants will place one hand on the chest and another on the sand bag placed over abdomen. This sand bag weighing 3-5 Kgs will provide resistance to breathing. These exercises will be performed in supine position. We will adjust the weight of the sandbag as per individual's level of 11-13 of 'Rating of Perceived Exercise (RPE)'.
  Supervised breathing exercises in two sets for 15 minutes with 5 minutes break between sets and 10 minutes rest after it will be performed
  Arms: Group B

SUMMARY:
This study is a randomised control trial and the purpose of this study is to determine the effects of core strengthening on trunk endurance after core strengthening with resistive versus non-resistive diaphragmatic training in lower cross syndrome.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of core strengthening on trunk endurance after core strengthening with resistive versus non-resistive diaphragmatic training in lower cross syndrome.

Core stability of young adults (age: 19-30 years) will be determined using McGill's muscular endurance test battery:

1. Flexor endurance test
2. Extensor endurance test
3. Right lateral endurance test
4. Left lateral endurance test Scores will be taken three times for each test; the average of each text will be noted for each participant.

Data collection procedure: Participants of interest would be approached and explained about the research. Informed written consent will be taken. Recruited participants will be allocated to either of the groups through a sealed opaque envelope method. McGill's Torso Muscular Endurance Test Battery will be used and baseline and post-intervention scores will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-30 years
* Both genders
* Positive modified Thomas test
* Positive prone hip extension strength test
* Positive trunk flexion strength test
* Tight erector spinae
* Asia pacific BMI normal and overweight (18.5-24.9 Kg/m2)
* Local intermittent lumbar pain
* Mild to moderate pain (NPRS 1-6)
* Painless movement and activity
* Pain only produced by sustained loading in relevant position, which is then relieved on moving from that posture

Exclusion Criteria:

* Shoulder pain
* Acute flare LBP
* Centralization and peripheralization of pain (21)
* Intermittent pain at limited end range (21)
* Leg symptoms when walking, eased in flexion (Signs of stenosis) (21)
* Pain due to repetitive movement (21)
* Paresthesia/numbness (21)
* Structural deformity (Kyphosis, lordosis, scoliosis, spondylosis, spondylolysis, spondylolisthesis)
* Curve reversal (21)
* Pregnancy
* Post surgery
* Degenerative and inflammatory spinal diseases

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in trunk flexor endurance test | 6 weeks
  Subject will sit on the test bench and place the upper body against a support with an angle of 60 ° from the test bed. The arms will be folded across the chest with the hands placed on the opposite shoulder. Subjects will be instructed to maintain the body position while the supporting wedge will be pulled back 10 cm to begin the test. The test will end when the upper body fell below the 60 ° angle.
Change in trunk extensor endurance test | 6 weeks
  Subjects will be laid prone with the lower body fixed to the test bed at the ankles, knees, and hips and the upper body extended. Subjects will rest their upper bodies on the floor before the exertion. At the beginning of the exertion, the upper limbs will be held across the chest with the hands resting on the opposite shoulders, and the upper body will be lifted off the floor until the upper torso is horizontal to the floor. Subjects will be instructed to maintain the horizontal position as long as possible.
Left lateral endurance test | 6 weeks
  The participants will assume a side-lying position with their legs fully extended and feet aligned on top of each other. Upon readiness, they will be instructed to transition into a full side-bridge position, ensuring that both legs remain extended and the sides of the feet are in contact with the floor. Timing will commence as they successfully maintain this position. The test will conclude if there is any noticeable change in the alignment of the participant's trunk. This test will be conducted twice with a 2-minute rest between intervals. The average duration of the two tests will be recorded on the participant's record sheet. The test will then
Right lateral endurance test | 6 weeks
  The participants will assume a side-lying position with their legs fully extended and feet aligned on top of each other. Their lower arm will be positioned under their body while the upper arm rests at their side. Upon readiness, they will be instructed to transition into a full side-bridge position, ensuring that both legs remain extended and the sides of the feet are in contact with the floor. Timing will commence as they successfully maintain this position. The test will conclude if there is any noticeable change in the alignment of the participant's trunk. This test will be conducted twice with a 2-minute rest between intervals. The average duration of the two tests will be recorded on the participant's record sheet. The test will then

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan